CLINICAL TRIAL: NCT03001063
Title: Mental Health in Adults and Children: Frugal Innovations
Brief Title: Mental Health in Adults and Children- Frugal Innovations (MAC-FI): Adult Depression Component
Acronym: MAC-FI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Simon Fraser University (Other)
Collaborators: Grand Challenges Canada (Other); Ministry of Labour - Invalids and Social Affairs (Unknown)
Responsible Party: Principal Investigator, John O'Neil, Dean, Faculty of Health Sciences, Simon Fraser University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0762-05
Record Dates: First submitted 2016-12-20; First posted 2016-12-22 (Estimated); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): This arm will receive the Supported Self- Management intervention, which consists of bibliotherapy that is provided with the regular support of health or social workers for a duration of two months.
  Interventions: Other: Supported Self-Management
- Control (Other): This arm will receive enhanced treatment as usual, which consists of a leaflet with information about depression and regular care as provided by primary care centres. The control arm will receive the intervention after the intervention arm has completed the intervention period.
  Interventions: Other: Enhanced treatment as usual

INTERVENTIONS:
Other: Supported Self-Management — This Supported Self-Management intervention consists of bibliotherapy (the Antidepressant Skills Workshop) that is provided to a patient by a health or social worker. The patient is supported in the use of the skills found in the workbook over the course of two months. The skills in the workbook are based on the principles of Cognitive Behavioural Therapy.
  Arms: Intervention
Other: Enhanced treatment as usual — Participants in the control arm will received enhanced treatment as usual in the form of usual care at primary care centres and a leaflet providing information about depression.
  Arms: Control

SUMMARY:
This stepped wedge, randomized controlled trial will test the effectiveness of a Supported Self-Management intervention for depression among adults in Vietnam. The intervention will be delivered at the community level in 8 Vietnamese provinces by primary care providers and social workers. The intervention group will receive the Supported Self-Management intervention, while the control group will receive enhanced treatment as usual. The primary outcome measure for depression is the Self-Reporting Questionnaire-20 (SRQ-20). The World Health Organization's Disability Assessment Scale (WHODAS 2.00 and the CAGE (Concern/Cut-down, Anger, Guilt, and Eye-opener) measures are also used to assess functional ability and alcohol misuse.

ELIGIBILITY:
Inclusion Criteria:

* Score of >7 on SRQ-20 indicating depression caseness
* Consent to participate and complete all measures

Exclusion Criteria:

* Cognitive disturbance
* Psychotic symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 376 (Actual)
Dates: Start 2016-03; Primary Completion 2019-01 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Self-Reporting Questionnaire 20 (SRQ-20) | Two months

SECONDARY OUTCOMES:
World Health Organization's Disability Assessment Scale (WHODAS 2.0) | Two months

CONTACTS AND LOCATIONS:
Overall Officials: John O'Neil, PhD, Principal Investigator — Simon Fraser University; Vu Cong Nguyen, MD, Principal Investigator — Institute of Population, Health and Development
Locations (1):
- Institute of Population, Health and Development, Hanoi, Vietnam

REFERENCES:
- [Derived] Murphy JK, Xie H, Nguyen VC, Chau LW, Oanh PT, Nhu TK, O'Neil J, Goldsmith CH, Van Hoi N, Ma Y, Lou H, Jones W, Minas H. Is supported self-management for depression effective for adults in community-based settings in Vietnam?: a modified stepped-wedge cluster randomized controlled trial. Int J Ment Health Syst. 2020 Feb 12;14:8. doi: 10.1186/s13033-020-00342-1. eCollection 2020. PMID 32071614
- [Derived] Murphy J, Goldsmith CH, Jones W, Oanh PT, Nguyen VC. The effectiveness of a Supported Self-management task-shifting intervention for adult depression in Vietnam communities: study protocol for a randomized controlled trial. Trials. 2017 May 5;18(1):209. doi: 10.1186/s13063-017-1924-5. PMID 28476148